CLINICAL TRIAL: NCT05912608
Title: Searching Optimal Tailored Strategy for Repair of Acute Type A Acute Aortic Dissection
Brief Title: Optimal Strategy for Repair of Type A Acute Aortic Dissection
Acronym: TARAD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Cardiologique du Nord (Other)
Collaborators: Henri Mondor University Hospital (Other); Universita degli Studi di Genova (Other); Pitié-Salpêtrière Hospital (Other); Ospedale San Camillo, Rome, Italy (Unknown)
Responsible Party: Principal Investigator, Francesco Nappi, Director, Centre Cardiologique du Nord
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN-202201173-1; CN-202201173-1 (Registry Identifier: TAAD)
Record Dates: First submitted 2023-05-28; First posted 2023-06-22 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Aortic Dissection
Keywords: Type A Acute Aortic Dissection (TAAAD); Root-Sparing Replacement; Hemiarch Procedures; Ascending Aorta Replacement; Total Arch Replacement (TARP); Frozen Elephant Trunk (FET)
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative Type A Acute Aortic Dissection Repair (TAAAD-R) (Active Comparator): All conservative TAAAD-R will be performed through a median sternotomy. The conservative TAAAD-R will include patients receiving valve-sparing root procedures and recipients of ascending aortic root sparing replacement if the intima separation extended into the sinuses resulting in commissural collapse.When necessary, the hemiarch technique will be used with a limited extension of the conservative procedure by resection of all the aortic tissue up to the left common carotid artery and which will be dictated according to the presentation of the lesion.
  Interventions: Procedure: Conservative TAAAD-R; Procedure: Extensive TAAAD-R
- Extensive Type A Acute Aortic Dissection Repair (TAAAD-R) (Other): All extensive TAAAD-R will be performed through a median sternotomy.The extensive TAAAD-R will include patients receiving replacement of the aortic root and total arch replacement procedures (TARP)
  Interventions: Procedure: Conservative TAAAD-R; Procedure: Extensive TAAAD-R

INTERVENTIONS:
Procedure: Conservative TAAAD-R — Cardiac arrest will be ensured using antegrade potassium-rich cardioplegia solution delivered directly into the coronary ostium or after coronary sinus cannula insertion, in patients with aortic regurgitation aorta will be resected down to the sinotubular junction and the thrombus located in the false lumen of the aortic root will be removed so that the aortic lesion could be visualized. The commissures will be resuspended using 4-0 or 5-0 sutures reinforced with a Teflon pledget over each commissure. A 4-0 or 5-0 polypropylene suture will be chosen to seal the proximal anastomosis and this suture line will also be used to secure the intima to the adventitia. In patients revealing normal-sized aortic roots associated with poor-quality valve leaflets, concomitant aortic valve replacement with conventional xenograft or mechanical prosthesis will be preferred.
  Other Names: Ascending aortic root sparing replacement with or without hemiarch repair
Procedure: Extensive TAAAD-R — Patients who experienced dilatation of the sinuses of Valsalva >4.5 cm in diameter on computed tomography imaging, those with connective tissue disease, or those in whom intimal tears extended into the sinuses, will undergoing replacement of the aortic root using a biologic or mechanical composite valve graft or valve-sparing root reimplantation procedure.Total arch replacement procedures (TARP) will fulfilled with the use of deep hypothermic circulatory arrest and with either antegrade or retrograde cerebral perfusion, maintaining systemic cooling between 19°C to 25°C and depending on the surgeon's practice.TARPs will be carried out using 1- and 4-branch grafts and involved the resection of all the aortic tissue up to the left common carotid artery (total hemiarch) or reimplantation of the innominate trunk only (partial hemiarch).
  Other Names: Aortic root procedures.TARP procedures

SUMMARY:
Acute type A aortic dissection (TAAD) persists as a clinicopathologic entity with high lethality in the current era. Several procedures are presently used to repair the TAAAD. The objective of this study is to analyze two groups of individuals using a conservative approach through root-sparing and hemiarch techniques in patients who are hospitalized in higher-risk clinical conditions or more aggressive procedures such as root replacement and total arch replacement in low-risk patients.

DETAILED DESCRIPTION:
The target population enrolled in the registry includes patients with TAAAD.The high volume of patients that will be enrolled in this registry will receive proximal and distal aortic repair in elective, urgent or emergency clinical condition. Efforts of investigators will be concentrated in TAAAD repair using a conservative approach of root preservation and hemiarch reconstruction in the majority of patients who will be referred in critical clinical condition. High-risk patients with older age or more comorbidities had more conservative repairs to limit surgical insult to these complicated patients. Total arch reconstruction and root replacement will be optional procedures for specific subgroups of patients who may benefit from a more complex index finger operation without incurring additional immediate risk.

Investigators hope to demonstrate a reduction in operative mortality and an improvement in early and late outcomes. The experience of investigators will be summarized in an algorithm for TAAAD repair with an analysis of early morbidity and mortality, as well as late survival and no reoperation.

ELIGIBILITY:
Inclusion Criteria:

* TAAD or intramural hematoma involving the ascending aorta
* Patients aged > 18 years
* Symptoms started within 7 days from surgery
* Primary surgical repair of acute TAAD
* Any other major cardiac surgical procedure concomitant with surgery for TAAD.

Exclusion Criteria:

* Patients aged < 18 years
* Onset of symptoms > 7 days from surgery
* Prior procedure for TAAD
* Concomitant endocarditis;
* TAAD secondary to blunt or penetrating chest trauma.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Operative Mortality (OM) | 30-day
  Patients who died within 30 days
Rate of Transient Neurologic Deficit (TND) | 30-day
  Number of participants who will complicate postoperatively with episode of TND which will include complication rate such as confusion, delirium, agitation
Rate of permanent Neurologic Deficit (PND) | 30-day
  Number of participants with acute episode of a focal or global neurological deficit. Rates of alteration of degree of consciousness, hemiplegia, hemiparesis, numbness or sensory loss affecting one side of the body, dysphasia or aphasia, hemianopsia, amaurosis fugax. To consider rate of other neurologic signs or symptoms consistent with stroke duration of focal or global neurologic deficit greater than 24 hours.

SECONDARY OUTCOMES:
Rate of perioperative Myocardial Infarction (MI) | 30-day
  Number of participants with MI based on fourth universal definition.
Rate of spinal Cord Injury (SCI) | 30-day
  Number of participants with SCI intended as rate of paraplegia and/or paraparesis
Rate of composite of Major Adverse Events (MAE) | 30-day
  Number of participants with MAE which will include the composite rate of myocardial infarction, cerebrovascular accident, need for dialysis, or need for tracheostomy according to Common Terminology Criteria for Adverse Events v4.0 (CTCAE)
Rate of composite of Major Adverse Pulmonary Events (MAPE) | 30-day
  Number of participants with MAPE which will include the composite rate of intubation >48 hours, pneumonia, reintubation, tracheostomy according to the Common Terminology Criteria for Adverse Events v4.0 (CTCAE)
Rate of reintervention | 10 years
  The number of participants who will require reoperation for the aortic valve, proximal aorta, or distal aorta.
Late survival | 10 years
  The secondary endpoint of the study is the evaluation of late survival

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Nappi, Principal Investigator — Cardiac Surgery Centre Cardiologique du Nord de Saint-Denis, Paris, France
Locations (1):
- Francesco Nappi, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Biancari F, Juvonen T, Fiore A, Perrotti A, Herve A, Touma J, Pettinari M, Peterss S, Buech J, Dell'Aquila AM, Wisniewski K, Rukosujew A, Demal T, Conradi L, Pol M, Kacer P, Onorati F, Rossetti C, Vendramin I, Piani D, Rinaldi M, Ferrante L, Quintana E, Pruna-Guillen R, Rodriguez Lega J, Pinto AG, Acharya M, El-Dean Z, Field M, Harky A, Nappi F, Gerelli S, Di Perna D, Gatti G, Mazzaro E, Rosato S, Raivio P, Jormalainen M, Mariscalco G. Current Outcome after Surgery for Type A Aortic Dissection. Ann Surg. 2023 Oct 1;278(4):e885-e892. doi: 10.1097/SLA.0000000000005840. Epub 2023 Mar 13. PMID 36912033
- [Result] Benedetto U, Dimagli A, Kaura A, Sinha S, Mariscalco G, Krasopoulos G, Moorjani N, Field M, Uday T, Kendal S, Cooper G, Uppal R, Bilal H, Mascaro J, Goodwin A, Angelini G, Tsang G, Akowuah E. Determinants of outcomes following surgery for type A acute aortic dissection: the UK National Adult Cardiac Surgical Audit. Eur Heart J. 2021 Dec 28;43(1):44-52. doi: 10.1093/eurheartj/ehab586. PMID 34468733
- [Result] Geirsson A, Shioda K, Olsson C, Ahlsson A, Gunn J, Hansson EC, Hjortdal V, Jeppsson A, Mennander A, Wickbom A, Zindovic I, Gudbjartsson T. Differential outcomes of open and clamp-on distal anastomosis techniques in acute type A aortic dissection. J Thorac Cardiovasc Surg. 2019 May;157(5):1750-1758. doi: 10.1016/j.jtcvs.2018.09.020. Epub 2018 Sep 29. PMID 30401530
- [Result] Harris KM, Nienaber CA, Peterson MD, Woznicki EM, Braverman AC, Trimarchi S, Myrmel T, Pyeritz R, Hutchison S, Strauss C, Ehrlich MP, Gleason TG, Korach A, Montgomery DG, Isselbacher EM, Eagle KA. Early Mortality in Type A Acute Aortic Dissection: Insights From the International Registry of Acute Aortic Dissection. JAMA Cardiol. 2022 Oct 1;7(10):1009-1015. doi: 10.1001/jamacardio.2022.2718. PMID 36001309
- [Result] Czerny M, Schoenhoff F, Etz C, Englberger L, Khaladj N, Zierer A, Weigang E, Hoffmann I, Blettner M, Carrel TP. The Impact of Pre-Operative Malperfusion on Outcome in Acute Type A Aortic Dissection: Results From the GERAADA Registry. J Am Coll Cardiol. 2015 Jun 23;65(24):2628-2635. doi: 10.1016/j.jacc.2015.04.030. PMID 26088302
- [Result] O'Hara D, McLarty A, Sun E, Itagaki S, Tannous H, Chu D, Egorova N, Chikwe J. Type-A Aortic Dissection and Cerebral Perfusion: The Society of Thoracic Surgeons Database Analysis. Ann Thorac Surg. 2020 Nov;110(5):1461-1467. doi: 10.1016/j.athoracsur.2020.04.144. Epub 2020 Jun 26. PMID 32599034